CLINICAL TRIAL: NCT01742169
Title: Center for Advancing Equity in Clinical Preventive Services Project 1B: Improving Rates of Colorectal Cancer Screening Among Never Screened Patients
Brief Title: Improving Rates of Colorectal Cancer Screening Among Never Screened Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Baker, Chief, Division of General Internal Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 1P01HS021141-01-Project1B; 1P01HS021141-01 (NIH)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Cancer Screening; Fecal Occult Blood Testing
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Outreach and Reminder Intervention (Experimental): Participants randomized to this arm will receive the Outreach and Reminder intervention.
  Interventions: Behavioral: Outreach and Reminder Intervention
- Usual Care (No Intervention): Patients assigned to this arm will receive usual care.

INTERVENTIONS:
Behavioral: Outreach and Reminder Intervention — This intervention includes (1) phone calls and text messages to inform participants that they are due for colorectal cancer (CRC) screening (2) mailed fecal occult blood test (FOBT) to participants so they can perform the test conveniently at home and mail them to the clinic, avoiding the need for a visit (3) plain language information and instructions to support understanding of CRC and FOBT use (4) a CRC screening coordinator to contact those still failing to complete testing by telephone or text (5) a feedback loop to patients regarding test results.
  Arms: Outreach and Reminder Intervention

SUMMARY:
The United States Preventive Services Task Force (USPSTF) recommends colorectal cancer (CRC) screening using fecal occult blood test (FOBT), sigmoidoscopy, or colonoscopy, beginning at age 50 and continuing until age 75. Despite this recommendation, rates of CRC screening remain inadequate and large disparities exist. Screening rates are lower among Black and Hispanic populations, in areas with high poverty rates, among individuals with low education, and for those who utilize Medicaid or lack health insurance. This study will determine the effectiveness of a multifaceted intervention to increase the number of patients who have never been screened for CRC and are cared for at a community health center (CHC) that complete a fecal immunochemical test (FIT) within 6 months of randomization to an intervention group compared to patients in a usual care group. We believe that the proposed intervention will improve the CRC screening rate in a cost-effective and sustainable way, ultimately leading to a reduction in the high rate of CRC.

Aim 1: To conduct a randomized controlled trial to determine if a multifaceted intervention increases the proportion of patients who complete a FOBT within 6-months of randomization.

Hypothesis 1: Compared to usual care, the intervention will increase the proportion of never-screened patients who complete FOBT within 6 months of randomization.

Aim 2: Assess the costs of the intervention and the costs per additional initial screening compared to patients who receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 to 75
* No documentation of previous CRC screening (FOBT, flexible sigmoidoscopy, or colonoscopy)
* Preferred language English or Spanish
* 2 visits to Erie Family Health Center in the past 2 years

Exclusion Criteria:

* Any of the following:

  1. colonoscopy within 10 years
  2. flexible sigmoidoscopy within 5 years
  3. a clinician order or referral for FOBT prior to the due date (indicating concern for gastrointestinal bleeding)
  4. medical conditions suggesting CRC screening through FOBT may be inappropriate, including chronic diarrhea, inflammatory bowel disease, iron deficiency, previous colonic polyp, use of medications in the previous 1 month that elevate the risk of a false-positive FOBT (i.e., plavix or warfarin), and medical conditions that make CRC screening inappropriate (metastatic cancer or previous total colectomy)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Completion of fecal occult blood test (FOBT) | Within 6 months of randomization to the intervention or control group
  This outcome will be assessed by querying the electronic health record (EHR) for all intervention and control patients to determine if an FOBT screening test was completed the community health center or documentation in the EHR that screening was completed elsewhere.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States